CLINICAL TRIAL: NCT05451693
Title: Outreach-ER: A Dementia Care Intervention Program
Status: Terminated | Type: Observational
Why Stopped: Planned recruitment was not feasible.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A22-086
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2022-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outreach-ER: Outreach-ER is a psychosocial intervention designed by dementia experts in the field of care partner interventions. The care plan will be personalized to the needs of the care partner/people living with dementia (PLWD).
  Interventions: Behavioral: Outreach-ER

INTERVENTIONS:
Behavioral: Outreach-ER — The intervention is similar to other care intervention/support programs such as REACH or New York University Caregiver Intervention (NYCUI). The Intervention is designed to be delivered over phone/virtual and in-home and will be conducted by Amplio, LLC consultants.

SUMMARY:
This is a feasibility/pilot, prospective cohort study to determine how to implement and refine Outreach-ER intervention for a larger clinical study. A key feature of Outreach-ER is to reach out to people living with dementia (PLWD) and their families following an emergency room visit or hospitalization. The outcome of this study will help in the overall goal of studying the impact of Outreach-ER in a larger clinical study and focus on outcomes relevant to PLWD and their care partners.

ELIGIBILITY:
Inclusion Criteria:

* PLWD with a recent Emergency department visit or admission at Regions Hospital
* Diagnosis of dementia based on international classification of diseases (ICD) Codes in the medical record
* Provides informed consent prior to participation
* Must be able to read and speak English
* PLWD Living at Home
* Age >=18 years for PLWD and their care partner

Exclusion Criteria:

* PLWD living in a nursing home/Long term care - Assisted living facility
* Current involvement in another clinical research study/trial for care partners
* PLWD medical record number (MRN) on the HealthPartners (HP) exclusion list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population includes people living with dementia (PLWD) who are treated at the Regions Hospital Emergency Department in Saint Paul, MN.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Neuroscience Research; Leah R Hanson, PhD, Principal Investigator — HealthPartners Neuroscience Research
Locations (2):
- United States (2):
  - Regions Hospital, Saint Paul, Minnesota
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 PLWD 4 Caregivers of PLWD
Groups:
- Outreach-ER (People Living With Dementia): Outreach-ER is a psychosocial intervention designed by dementia experts in the field of care partner interventions. The care plan will be personalized to the needs of the care partner/PLWD.
  Outreach-ER: The intervention is similar to other care intervention/support programs such as REACH or New York University Caregiver Intervention (NYCUI). The Intervention is designed to be delivered over phone/virtual and in-home and will be conducted by Amplio, LLC consultants.
- Outreach-ER (Caregiver): Caregiver to the PLWD also participating in the Outreach-ER program.
Period: Overall Study
Arm/Group | Outreach-ER (People Living With Dementia) | Outreach-ER (Caregiver)
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Outreach-ER (Caregivers of PLWD): Caregivers of PLWD also participating in the Outreach-ER program.
- Total: Total of all reporting groups
Arm/Group | Outreach-ER (People Living With Dementia) | Outreach-ER (Caregivers of PLWD) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9.8) | 65 (4.7) | 66.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Dementia Type [Count of Participants; unit: Participants]
  Late Onset Alzheimer's Disease | 2 | 0 | 2
  Lewy Body Dementia (Mixed) | 1 | 0 | 1
  Alzheimer's Disease with Down Syndrome | 1 | 0 | 1
  No Dementia | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempted Recruits for Feasibility and Acceptability of Outreach-ER
Description: Number of potential participant/care partner dyads contacted. Higher number indicates higher number of attempts as recruitment.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Outreach-ER: Outreach-ER is a psychosocial intervention designed by dementia experts in the field of care partner interventions. The care plan will be personalized to the needs of the care partner/PLWD.
  Outreach-ER: The intervention is similar to other care intervention/support programs such as REACH or New York University Caregiver Intervention (NYCUI). The Intervention is designed to be delivered over phone/virtual and in-home and will be conducted by Amplio, LLC consultants.
Arm/Group | Outreach-ER
Number analyzed (Participants) | 32
Participants | 32

2. Primary Outcome: Recruitment Rate for Feasibility and Acceptability of Outreach-ER
Description: Percentage of participant/care partner dyads who enroll and consent [range: 0-100%]. Higher number indicates more feasibility.
Time Frame: 4 months
Measure: Number; unit: percentage of attempted recruits
Arm/Group | Outreach-ER
Number analyzed (Participants) | 32
percentage of attempted recruits | 13

3. Primary Outcome: Participant Rate for Feasibility and Acceptability of Outreach-ER
Description: Percentage of participant/care partner dyads who start Outreach-ER program [range: 0-100%]. Higher number indicates more feasibility.
Time Frame: First day of intervention
Measure: Number; unit: percentage of attempted recruits
Arm/Group | Outreach-ER
Number analyzed (Participants) | 32
percentage of attempted recruits | 13

4. Primary Outcome: Completion Rate for Feasibility and Acceptability of Outreach-ER
Description: Percentage of participant/care partner dyads who complete intervention (7 or more visits) [range: 0-100%]. Higher number indicates more feasibility.
Time Frame: about 4 months
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Outreach-ER
Number analyzed (Participants) | 4
percentage of enrolled participants | 75

5. Primary Outcome: Session Specific Completion Rate for Feasibility and Acceptability of Outreach-ER
Description: Percentage of participant/care partner dyads who complete each intervention visit [range: 0-100%].
  Number of total intervention visits completed = total completed visits for the 4 dyads.
  Number of total intervention visits available = 6 visits x 4 dyads = 24 visits. Number of total intervention visits completed/24 total intervention visits x 100 = percentage.
  Higher number indicates more feasibility.
Time Frame: about 4 months
Measure: Number; unit: percentage of sessions completed
Units Other Than Participants: sessions
Arm/Group | Outreach-ER
Number analyzed (Participants) | 4
Number analyzed (sessions) | 24
percentage of sessions completed | 86

6. Primary Outcome: Questionnaire Specific Response Rate for Feasibility and Acceptability of Outreach-ER
Description: Percentage of participant/care partner dyads who complete each questionnaire [range: 0-100%].
  Number of total questionnaires completed = total completed questionnaires for the 4 dyads.
  Number of total questionnaires available = 3 questionnaires x 4 dyads x 2 visit time points = 24 available questionnaires.
  Number of total questionnaires completed/24 total questionnaires available x 100 = percentage.
  Higher number indicates more feasibility.
Time Frame: about 4 months
Measure: Number; unit: percentage of completed questionnaires
Units Other Than Participants: questionnaires
Arm/Group | Outreach-ER
Number analyzed (Participants) | 4
Number analyzed (questionnaires) | 24
percentage of completed questionnaires | 67

7. Secondary Outcome: Completeness of Specific Measures for Feasibility and Acceptability of Outreach-ER
Description: Percentage of care partners that respond to all of the items on each scale [range: 0-100%]. Higher number indicates more feasibility.
Time Frame: about 4 months
Measure: Number; unit: percentage of completed questions
Arm/Group | Outreach-ER
Number analyzed (Participants) | 4
percentage of completed questions | 75

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Outreach-ER (People Living With Dementia) | Outreach-ER (Caregivers of PLWD)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05451693/Prot_SAP_000.pdf